CLINICAL TRIAL: NCT02466776
Title: Comparison of Staples Versus Subcuticular Suture in Class III Obese Women Undergoing Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MemorialCare Health System (Other)
Collaborators: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Jennifer McNulty, MD, Maternal Fetal Medicine Specialist, MemorialCare Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 459-14
Record Dates: First submitted 2015-06-03; First posted 2015-06-09 (Estimated); Results first posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Obesity, Severe; Cesarean Section
MeSH Terms: conditions — Obesity, Morbid | interventions — Sutures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stainless steel staples (Active Comparator): Patients in this arm will receive stainless steel staples for skin closure at time of cesarean delivery (CD).
  Interventions: Device: Stainless steel staples
- Absorbable subcuticular Suture (Active Comparator): Patients will receive absorbable subcuticular suture for skin closure at time of cesarean delivery (CD).
  Interventions: Device: Absorbable subcuticular suture

INTERVENTIONS:
Device: Absorbable subcuticular suture — Patients will receive absorbable subcuticular suture for skin closure at time of cesarean delivery (CD).
  Other Names: 3-0 monocryl
  Arms: Absorbable subcuticular Suture
Device: Stainless steel staples — Patients will receive stainless steel staples for skin closure at time of cesarean delivery (CD).
  Other Names: Staples
  Arms: Stainless steel staples

SUMMARY:
The purpose of this study is to determine the optimal skin closure technique (staples versus subcuticular suture) at the time of cesarean delivery in Class III obese women with body mass index (BMI) of >/= 40kg/m2.

DETAILED DESCRIPTION:
A. To assess the rate of wound complications with staples versus subcuticular suture closure in women with a BMI of ≥ 40 kg/m2 undergoing cesarean delivery (CD).

B. No difference was observed in wound complication rates between staples and subcuticular suture skin closure in women with a BMI ≥ 40 kg/m2 undergoing cesarean delivery (CD).

C. At this time, optimal skin closure method in obese women with BMI ≥ 40 kg/m2 undergoing cesarean delivery remains unknown. More work is needed in this area to help reduce the complication rate in this very high-risk population.

ELIGIBILITY:
Inclusion Criteria:

1. Women > 18 years old undergoing cesarean delivery (CD)
2. BMI of >/= 40 kg/m2 as determined by height and weight reported during their admission
3. Live gestation 23 weeks or greater
4. Women who are able to follow-up 7-14 days after hospital discharge for a visual wound check.

Exclusion Criteria:

1. Active lupus flare
2. HIV/AIDS
3. Current treatment for cancer or h/o radiation to the abdomen/pelvis
4. Hypersensitivity to steri-strips

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer McNulty, MD, Principal Investigator — MemoriaCare HealthSystem
Locations (4):
- United States (4):
  - Long Beach Memorial Care Center for Women at Miller Children's Hospital Long Beach and Long Beach Memorial Hospital, Long Beach, California
  - Long Beach Memorial Care Center for Women at Miller Children's Hospital Long Beach, Long Beach, California
  - Long Beach Memorial Care Center, Long Beach, California
  - University of California, Irvine, Orange, California

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Stainless Steel Staples | Absorbable Subcuticular Suture
Started | 119 | 119
Completed | 119 | 119
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Absorbable Subcuticular Suture | Stainless Steel Staples | Total
Number analyzed (Participants) | 119 | 119 | 238
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.1 (5.6) | 31.4 (5.3) | 31.25 (0.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 119 | 238
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  African American | 22 | 19 | 41
  Asian | 5 | 10 | 15
  Caucasian | 22 | 24 | 46
  Hispanic | 68 | 59 | 127
  Other | 2 | 7 | 9
Region of Enrollment [Number; unit: participants]
  United States | 119 | 119 | 238
Married/partner [Count of Participants; unit: Participants] | 69 | 66 | 135
College Graduate [Count of Participants; unit: Participants] | 23 | 21 | 44
Private Insurance [Count of Participants; unit: Participants] | 31 | 28 | 59
Singleton Gestation [Count of Participants; unit: Participants] | 111 | 114 | 225
Gestational age at delivery [Mean (Standard Deviation); unit: Weeks] | 38.8 (1.9) | 38.2 (2.5) | 38.5 (0)
Number of previous cesarean delivery (CD) [Count of Participants; unit: Participants]
  o | 45 | 42 | 87
  1 | 36 | 42 | 78
  2 or more | 38 | 35 | 73
Time since last cesarean delivery (CD) [Count of Participants; unit: Participants]
  No history of prior cesarean delivery (CD) | 45 | 42 | 87
  Within 5 years | 41 | 44 | 85
  More than 5 years | 33 | 33 | 66
Diabetes [Count of Participants; unit: Participants]
  None | 82 | 77 | 159
  Pre-gestational | 19 | 19 | 38
  Gestational | 18 | 23 | 41
Hypertensive Disease [Count of Participants; unit: Participants]
  None | 85 | 73 | 158
  Pre-gestational | 9 | 16 | 25
  Gestational | 12 | 10 | 22
  Preeclampsia | 13 | 20 | 33
Tobacco use [Count of Participants; unit: Participants]
  None | 96 | 90 | 186
  Current | 7 | 3 | 10
  Past | 16 | 26 | 42
Chorioamnionitis [Count of Participants; unit: Participants] | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Composite Wound Complication at Hospital Discharge and 2 Weeks Postpartum
Description: Rate of wound complications defined as composite wound complication, which includes infection requiring antibiotics, hematoma, seroma, separation or disruption, and/or readmission to the hospital for wound concerns.
Time Frame: At hospital discharge, at 2 weeks postpartum and at 6 weeks postpartum
Population: The last 2 rows show the rate of healed versus non-healed wound complications out of the total number of wound complications diagnosed in the staples group (n=8) and suture group (n=5).
Measure: Count of Participants; unit: Participants
Groups:
- Stainless Steel Staples at HOSPITAL DISCHARGE; Stainless Steel Staples at 2 WEEKS POSTPARTUM; Stainless Steel Staples TOTAL WOUND COMPLICATIONS: Patients in this arm will receive stainless steel staples for skin closure at time of cesarean section.
  Stainless steel staples: Patients will receive stainless steel staples for skin closure at time of cesarean section.
- Absorbable Subcuticular Suture at HOSPITAL DISCHARGE; Absorbable Subcuticular Suture at 2 WEEKS POSTPARTUM; Absorbable Subcuticular Suture TOTAL WOUND COMPLCATIONS: Patients will receive absorbable subcuticular suture for skin closure at time of cesarean section.
  Absorbable subcuticular suture: Patients will receive absorbable subcuticular suture for skin closure at time of cesarean section.
Arm/Group | Stainless Steel Staples at HOSPITAL DISCHARGE | Absorbable Subcuticular Suture at HOSPITAL DISCHARGE | Stainless Steel Staples at 2 WEEKS POSTPARTUM | Absorbable Subcuticular Suture at 2 WEEKS POSTPARTUM | Stainless Steel Staples TOTAL WOUND COMPLICATIONS | Absorbable Subcuticular Suture TOTAL WOUND COMPLCATIONS
Number analyzed (Participants) | 118 | 119 | 119 | 119 | 119 | 119
Participants
  Composite wound complication | 8 | 5 | 15 | 16 | 23 | 21
  Infection | 0 | 0 | 3 | 2 | 3 | 2
  Superficial separation | 7 | 3 | 11 | 11 | 15 | 14
  Deep separation | 1 | 2 | 3 | 0 | 4 | 2
  Infection and separation | 0 | 0 | 1 | 3 | 1 | 3
  Healed at 6 weeks: number analyzed (Participants) | 8 | 5 | 15 | 12 | 0 | 0
  Healed at 6 weeks | 6 | 4 | 12 | 11 |  |
  Not healed at 6 weeks: number analyzed (Participants) | 8 | 5 | 15 | 12 | 0 | 0
  Not healed at 6 weeks | 2 | 1 | 3 | 1 |  |

2. Secondary Outcome: Number of Participants According to Skin Incision
Description: Date were analyzed with independent t, X2 and Fisher's exact tests, where applicable
Time Frame: At time of surgery and hospitalization
Measure: Count of Participants; unit: Participants
Arm/Group | Absorbable Subcuticular Suture | Stainless Steel Staples
Number analyzed (Participants) | 119 | 119
Participants
  Skin incision: Pfannenstiel | 114 | 118
  Skin incision: Midline vertical | 5 | 1

3. Secondary Outcome: Operating Surgeon Level
Description: Date were analyzed with independent t, X2 and Fisher's exact tests, where applicable
Time Frame: At time of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Stainless Steel Staples | Absorbable Subcuticular Suture
Number analyzed (Participants) | 119 | 119
Participants
  Surgeon level: Attending/Fellow | 67 | 66
  Surgeon level: Resident | 52 | 53

4. Secondary Outcome: Surgical Assistant Level
Description: Date were analyzed with independent t, X2 and Fisher's exact tests, where applicable
Time Frame: At time of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Stainless Steel Staples | Absorbable Subcuticular Suture
Number analyzed (Participants) | 119 | 119
Participants
  Assistant Level: Attending/Fellow | 101 | 97
  Assistant Level: Resident | 18 | 22

5. Secondary Outcome: Total Operative Time
Description: Date were analyzed with independent t, X2 and Fisher's exact tests, where applicable
Time Frame: At time of surgery and hospitalization
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Stainless Steel Staples: Patients in this arm will receive stainless steel staples for skin closure at time of cesarean section.
  Stainless steel staples: Patients will receive stainless steel staples for skin closure at time of cesarean delivery (CD).
- Absorbable Subcuticular Suture: Patients will receive absorbable subcuticular suture for skin closure at time of cesarean section.
  Absorbable subcuticular suture: Patients will receive absorbable subcuticular suture for skin closure at time of cesarean delivery (CD).
Arm/Group | Stainless Steel Staples | Absorbable Subcuticular Suture
Number analyzed (Participants) | 119 | 119
minutes | 43.4 (21.9) | 55.8 (26)

6. Secondary Outcome: Total Blood Loss
Description: Date were analyzed with independent t, X2 and Fisher's exact tests, where applicable
Time Frame: At time of surgery
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Stainless Steel Staples | Absorbable Subcuticular Suture
Number analyzed (Participants) | 119 | 119
mL | 773 (432) | 837 (447)

7. Secondary Outcome: Number of Participants With Blood Transfusion
Description: Date were analyzed with independent t, X2 and Fisher's exact tests, where applicable
Time Frame: At time of surgery and hospitalization
Measure: Count of Participants; unit: Participants
Arm/Group | Stainless Steel Staples | Absorbable Subcuticular Suture
Number analyzed (Participants) | 119 | 119
Participants | 4 | 8

8. Secondary Outcome: Change in Hemoglobin (Pre-delivery and Post-delivery)
Description: Date were analyzed with independent t, X2 and Fisher's exact tests, where applicable
Time Frame: At time of surgery (pre-delivery) and post-delivery
Measure: Mean (Standard Deviation); unit: Change in grams of hemoglobin
Arm/Group | Stainless Steel Staples | Absorbable Subcuticular Suture
Number analyzed (Participants) | 119 | 119
Change in grams of hemoglobin | 1.68 (1.5) | 1.93 (1.4)

9. Secondary Outcome: Neonatal Birthweight
Description: Date were analyzed with independent t, X2 and Fisher's exact tests, where applicable
Time Frame: At time of delivery
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Stainless Steel Staples | Absorbable Subcuticular Suture
Number analyzed (Participants) | 119 | 119
grams | 3406 (878) | 3426 (711)

10. Secondary Outcome: Number of Participants With 5 Minute Apgar Score <7
Description: Date were analyzed with independent t, X2 and Fisher's exact tests, where applicable The Apgar score, developed by Virginia Apgar describes the condition of the newborn infant immediately after birth and, when properly applied, is a tool for standardized assessment 18. It also provides a mechanism to record fetal-to-neonatal transition. This scoring system provided a standardized assessment for infants after delivery. The Apgar score comprises five components: 1) color, 2) heart rate, 3) reflexes, 4) muscle tone, and 5) respiration, each of which is given a score of 0, 1, or 2. The Apgar score ranges from 0 (lowest, poor outcome) to 10 (highest, good outcome).
Time Frame: At time of delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Stainless Steel Staples | Absorbable Subcuticular Suture
Number analyzed (Participants) | 119 | 119
Participants | 2 | 1

11. Secondary Outcome: Number of Participants Receiving Postpartum Prophylactic Anticoagulation
Description: Date were analyzed with independent t, X2 and Fisher's exact tests, where applicable
Time Frame: During hospitalization
Measure: Count of Participants; unit: Participants
Arm/Group | Stainless Steel Staples | Absorbable Subcuticular Suture
Number analyzed (Participants) | 119 | 119
Participants | 66 | 74

12. Secondary Outcome: Total Length of Hospital Stay
Description: Date were analyzed with independent t, X2 and Fisher's exact tests, where applicable
Time Frame: At time of surgery and hospitalization
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Stainless Steel Staples | Absorbable Subcuticular Suture
Number analyzed (Participants) | 119 | 119
days | 4.9 (0.9) | 4.9 (2.1)

13. Secondary Outcome: Patient Pain Score (From 1 to 10)
Description: Patients' pain associated with their wound within 7-14 days after hospital discharge using a self-administered questionnaire that asked patients to rate their pain on a scale of 0 (no pain) to 10 (worst pain).
Time Frame: Within 2 weeks postpartum
Measure: Median (95% Confidence Interval); unit: Score on a scale
Arm/Group | Absorbable Subcuticular Suture | Stainless Steel Staples
Number analyzed (Participants) | 113 | 114
Score on a scale | 2 [1 to 3] | 2 [1 to 3]

14. Secondary Outcome: Patient Satisfaction With Wound Healing and Appearance
Description: Patients' satisfaction with the healing of their wound within 7-14 days after hospital discharge using a self-administered questionnaire that asked patients to rate their overall satisfaction with their wound healing and appearance (1=least satisfied, 10=most satisfied). Patients were also asked to rate their concern regarding their wound healing (1= least concerned and 10 = most concerned).
Time Frame: At time of hospital discharge and at 2 weeks postpartum
Measure: Median (95% Confidence Interval); unit: Score on a scale
Groups:
- Absorbable Subcuticular Suture at HOSPITAL DISCHARGE: Patients will receive absorbable subcuticular suture for skin closure at time of cesarean delivery (CD).
  Absorbable subcuticular suture: Patients will receive absorbable subcuticular suture for skin closure at time of cesarean delivery (CD).
- Stainless Steel Staples at 2 WEEKS POSTPARTUM: Patients in this arm will receive stainless steel staples for skin closure at time of cesarean delivery (CD).
  Stainless steel staples: Patients will receive stainless steel staples for skin closure at time of cesarean delivery (CD).
Arm/Group | Absorbable Subcuticular Suture at HOSPITAL DISCHARGE | Stainless Steel Staples at 2 WEEKS POSTPARTUM
Number analyzed (Participants) | 113 | 114
Score on a scale
  Wound appearance satisfaction (1=least, 10=most) | 10 [9 to 10] | 10 [9 to 10]
  Concern about wound healing (1=least, 10=most) | 1 [1 to 2] | 1 [1 to 2]

ADVERSE EVENTS:
Groups:
- Stainless Steel Staples: Patients in this arm will receive stainless steel staples for skin closure at time of cesarean section.
  Stainless steel staples: Patients will receive stainless steel staples for skin closure at time of cesarean section.
- Absorbable Subcuticular Suture: Patients will receive absorbable subcuticular suture for skin closure at time of cesarean section.
  Absorbable subcuticular suture: Patients will receive absorbable subcuticular suture for skin closure at time of cesarean section.
Arm/Group | Stainless Steel Staples | Absorbable Subcuticular Suture
All-Cause Mortality (participants affected / at risk) | 0/119 | 0/119
Serious Adverse Events (participants affected / at risk) | 0/119 | 0/119
Other Adverse Events (participants affected / at risk) | 0/119 | 0/119

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes